CLINICAL TRIAL: NCT04693494
Title: Effectiveness of a Training Program for Parents of Babies in Their First Year of Life to Achieve Motor Milestones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Luis Fernandez, Physical Therapist, Universidad San Jorge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ufernandez2020
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Term; Healthy; Motor Delay; Development, Infant
Keywords: motor milestones; term; newborn; motor development
MeSH Terms: conditions — Psychomotor Disorders

STUDY DESIGN:
Intervention Model Description: Intervention and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded: spontaneous behavior of babies is evaluated, that doesn't depend of having knowledge of the intervention. Outcomes assessor doesn't know the evaluated baby group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Four training sessions (before the baby is 1 month old, at 3 months, at 6 and at 9 months old) teaching the main motor milestones to get in the next 3 months and how to help infants with the correct stimuli, positions or plays; triptychs containing the main points explained at the session and links to short videos about the given advices.
  Three evaluations of motor milestones at the age of 9, 12, and 15 months old
  Interventions: Other: Training program
- Control group (No Intervention): Three evaluations of motor milestones at the age of 9, 12, and 15 months old

INTERVENTIONS:
Other: Training program — Training program consisting in 4 sessions with information about milestones to achieve and advices for motor development. Triptychs and short videos containing the main points containing the main points.
  Arms: Intervention group

SUMMARY:
this study compares motor development of two groups of healthy term babies at the end of their first year of life. Parents of the intervention group have received a training program consisting in advices about correct positions, stimuli, how to play or how to carry their babies. The purpose of this study is to know if motor development can be improved by the environment.

DETAILED DESCRIPTION:
Infants in both groups are recruited by the principal investigator at the hospital within two to three days after birth. An initial assessment was carried out at 2 months of age.

Intervention group:

1. Four training sessions (before the baby is 1 month old, at 3 months, at 6, and at 9 months old) teaching the main motor milestones to get in the next 3 months and how to help infants with the correct stimuli, positions or plays; triptychs containing the main points explained at the session and links to short videos about the given bits of advice.
2. Three evaluations of motor milestones at 9, 12, and 15 months old.

Control group:

1. Three evaluations of motor milestones at 9, 12, and 15 months old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy-term infants
* Male and female
* Apgar score of at least 7 in the first minute and at five minutes.
* Natural or cesarean birth
* Absence of congenital malformations or orthopedic injury
* Absence of known congenital or genetic pathology
* Normal neurological medical examination of the newborn at hospital discharge.

Exclusion Criteria:

* Newborns who have required hospitalization before being enrolled.
* Multiple births

Ages: 1 Day to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Score of the Alberta Infant Motor Scale (AIMS) at month 9 | 9 months old
  AIMS is a validated observational scale for measurement of motor milestones. Higher scores mean a better outcome. Depending on the score, the percentile is obtained.
Score of the Alberta Infant Motor Scale (AIMS) at month 12 | 12 months old
  AIMS is a validated observational scale for measurement of motor milestones. Higher scores mean a better outcome. Depending on the score, the percentile is obtained.Depending on the score, the percentile is obtained.
Score of the Alberta Infant Motor Scale (AIMS) at month 15 | 15 months old
  AIMS is a validated observational scale for measurement of motor milestones. Higher scores mean a better outcome. Depending on the score, the percentile is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernández Sola, Physical Th, Principal Investigator — Universidad San Jorge; Beatriz Cano Díez, Physical Th, Study Director — Universidad San Pablo CEU
Locations (1):
- Universidad San Jorge, Zaragoza, Aragon, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD after deidentified
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years
Access Criteria: Información will be shared with editors or other investigators

REFERENCES:
- [Derived] Fernandez-Sola L, Cano-Diez B, Pons-Solaz Y, Vera-Egido B, Moreno-Gonzalez S. Effectiveness of a training program for the acquisition of motor milestones in infants: a randomized clinical trial. Ital J Pediatr. 2025 Jan 31;51(1):23. doi: 10.1186/s13052-025-01849-4. PMID 39891196